CLINICAL TRIAL: NCT05947266
Title: Intervening With Haitian Immigrants in the U.S. to Improve HIV Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMH34133481
Record Dates: First submitted 2023-06-26; First posted 2023-07-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV Infection Primary
Keywords: Viral suppression

STUDY DESIGN:
Intervention Model Description: Prospective, quasi-experimental, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haitian immigrant iENGAGE (H-iENGAGE) intervention (Experimental): 1. Enrollment;
  2. Baseline assessment;
  3. Upon baseline completion, scheduling of H-iENGAGE sessions 1 through 4
  4. Following Session 4, conduct Process evaluation;
  5. Post-intervention assessment;
  6. Six-month follow up assessment*
     *Six participants will complete AIM 3: Identify multi-level implementation factors contributing to intervention outcomes, using photovoice in mixed methods.
  7. End of study participation
  Interventions: Behavioral: an adaptation of the iENGAGE

INTERVENTIONS:
Behavioral: an adaptation of the iENGAGE — Haitian immigrant iENGAGE (H-iENGAGE) is an adaptation of the iENGAGE intervention culturally adapted for Haitian immigrants with HIV that will be tested in a quasi-experimental pilot for preliminary efficacy among recently diagnosed or nonvirally suppressed adults across two Federally Qualified Health Centers (FQHCs) in Miami.
  Other Names: Haitian immigrant iENGAGE (H-iENGAGE)

SUMMARY:
The goal of this clinical trial is to test a culturally tailored engagement and retention intervention for Haitian Immigrants Living With HIV (HILWH). The main questions it aims to answer are:

* Does this intervention result in measurable engagement and retention in care?
* Does this intervention result in measurable viral suppression within 6 months?

Participants will

* participate in a pilot health intervention entailing 4 individual meetings, approximately once monthly over a six-month period and completing research questionnaires at enrollment, post-intervention and at 6 months post-enrollment.
* Six participants who have completed the pilot intervention and agree to take part, will participate in the photovoice portion of the study. This activity will consist of 6 additional meetings where participants will be taught about using photographs to illustrate their experience participating in the study and take and display photographs.

DETAILED DESCRIPTION:
Research design: The proposed study will test a culturally tailored engagement and retention intervention for Haitian immigrants living with HIV (HILWH). This is sequential mixed-methods formative pilot research that is designed to examine engagement and retention in care, and viral suppression (VS) for HILWH and adapt a promising intervention that will result in viral suppression between baseline and a 6 month follow-up assessment. The pilot will be conducted as a prospective, quasi-experimental single arm with a sample of newly diagnosed or nonvirally suppressed HIWLH adults drawn from 2 Federally Qualified Health Centers (FQHC) sites in Miami.

Procedures to be used:

AIM 1 mixed methods (quantitative and qualitative) data collection on barriers and facilitators to viral suppression among HILWH. Quantitative questionnaires will be completed by health care service providers and HILWH who will also participate in a Focus group. A sample of HILWH will participate in individual in-depth interviews.

AIM 2 consists of a pilot health intervention entailing completing research questionnaires at enrollment, post-intervention and at 6 months post-enrollment. In addition, participants will have 4 individual meetings, approximately once monthly over a six month period.

AIM 3 Photovoice participants will be 6 participants who have completed the pilot intervention (AIM 2) and agree to participate in the photovoice portion of the study. This activity will consist of 6 additional meetings where participants will be taught about using photographs to illustrate their experience participating in the study and taking photographs. This activity is expected to take approximately 8 additional hours over 2 and a half months. For these six participants, the total amount of time will be approximately 20 hours over 8 and 1/2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Seropositive for HIV
2. Either a recent HIV diagnosis (within the last 2 months) or non-virally suppressed.
3. Migrated to the US from Haiti

Exclusion Criteria:

1. Virally suppressed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Care of Engagement Index Score | Baseline, post-intervention (week 12 to 14 post baseline), 6-month post-baseline follow up
  Change in Engagement in Care score over time, including comfort and communication with provider
Viral suppression | Baseline, 6-month post-baseline follow up
  Change in HIV load measurement toward a target of less than 200 copies/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Care Resource, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No